CLINICAL TRIAL: NCT06823037
Title: HAPPI (Hormonal Contraception Access Through Pharmacist Prescribing Implementation): Phase 2 (Aim 1)
Brief Title: Hormonal Contraception Access Through Pharmacist Prescribing Implementation
Acronym: HAPPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EMPOWERX INC (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Jenny Newlon, Research Director, EMPOWERX INC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R44DP006691 (NIH)
Record Dates: First submitted 2025-01-20; First posted 2025-02-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Contraception; Pharmaceutical Services; Access and Linkage to Healthcare; Technology Use
Keywords: community pharmacy; access to care; pharmacist services; birth control; health technology; scope of practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAPPI Pharmacies (Other): This is a single-arm trial, so all pharmacies will serve as their own control. We will enroll 15 community pharmacies. These 15 pharmacies will continue to provide birth control services as normal for several months (control). Then, we will introduce the intervention: the HAPPI software. The pharmacies will continue to provide birth control services while using the HAPPI software in place of any paper or electronic processes that they were previously using. The results will then be compared between the control and the intervention period.
  Interventions: Other: HAPPI software

INTERVENTIONS:
Other: HAPPI software — We will enroll 15 community pharmacies. These 15 pharmacies will continue to provide birth control services as normal for several months (control).
  Then, we will introduce the intervention: the HAPPI software. The pharmacies will continue to provide birth control services while using the HAPPI software in place of any paper or electronic processes that they were previously using. The results will then be compared between the control and the intervention period.

SUMMARY:
The goal of this clinical trial is to learn if use of the HAPPI software can improve pharmacist-provided birth control services. The main questions it aims to answer are:

1. Does the HAPPI software make it easier for pharmacists to provide birth control services in their pharmacy?
2. Does the HAPPI software make it easier for patients to access birth control?

Researchers will compare pharmacists' implementation and patients' access when using the HAPPI software and when not using the HAPPI software to see if the software improves implementation and access.

Participants will include pharmacists and patients. Pharmacists will be asked to provide birth control services as normal while using the HAPPI software. Patients will be asked to receive birth control services from a pharmacist as normal, while using the HAPPI software.

ELIGIBILITY:
PHARMACIST Participants

Inclusion Criteria:

* 18 years of age or older
* Provide birth control services in a participating pharmacy
* Use the HAPPI software to provide birth control services

Exclusion Criteria:

* None

PATIENT Participants

Inclusion Criteria:

* 18 years of age or older
* Seek birth control services at a participating pharmacy
* Use the HAPPI software to receive birth control services at a participating pharmacy

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Implementation - Service Characteristics Number of Pharmacists | up to 5 months
  Implementation outcomes will focus on how the service (pharmacist-prescribed contraceptive services) is implemented.
  Name of the Measurement: Implementation - Service Characteristics Measurement Tool: Pharmacy Service Characteristics Questionnaire
  Unit of Measure:
  * Number of pharmacists involved in providing birth control services
Implementation - Service Characteristics Number of Pharmacy Staff | up to 5 months
  Implementation outcomes will focus on how the service (pharmacist-prescribed contraceptive services) is implemented.
  Name of the Measurement: Implementation - Service Characteristics Measurement Tool: Pharmacy Service Characteristics Questionnaire
  Unit of Measure:
  * Number of pharmacy staff (non-pharmacists) involved in providing birth control services
Implementation - Service Characteristics Cash Pay | up to 5 months
  Implementation outcomes will focus on how the service (pharmacist-prescribed contraceptive services) is implemented.
  Name of the Measurement: Implementation - Service Characteristics Measurement Tool: Pharmacy Service Characteristics Questionnaire
  Unit of Measure:
  * Total amount of money coming in (revenue) from the service via cash pay
Implementation - Service Characteristics Insurance Billing | up to 5 months
  Implementation outcomes will focus on how the service (pharmacist-prescribed contraceptive services) is implemented.
  Name of the Measurement: Implementation - Service Characteristics Measurement Tool: Pharmacy Service Characteristics Questionnaire
  Unit of Measure:
  * Total amount of money coming in (revenue) from the service via insurance billing
Implementation - Proctor Implementation Outcomes | up to 5 months
  Implementation outcomes will be measured using Proctor et al.'s (2011) implementation framework. The domains in this framework include appropriateness, acceptability, adoption, feasibility, and fidelity. Survey items will map to each of these domains.
  Name of the measurement: Implementation - Proctor Implementation Outcomes Measurement tool: Implementation Outcomes Scale Unit of Measure: 5-point Likert-type scale (1= strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree). This same scale is used for all implementation domains (appropriateness, acceptability, adoption, feasibility, and fidelity).

SECONDARY OUTCOMES:
Access to Care | up to 5 months
  Access to Care outcomes will be assessed using a previously developed scale of Access to Contraceptive Care (Newlon 2021) that assesses patients' access in terms of approachability, acceptability, availability and accommodation, affordability, appropriateness, and privacy.
  Unite of measure: 5-point Likert-type scale (1= strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree). This same scale is used for all implementation domains (approachability, acceptability, availability and accommodation, affordability, appropriateness, and privacy).

CONTACTS AND LOCATIONS:
Locations (1):
- EmpoweRx, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Our clinical trial uses proprietary information related to the software that is the basis for our intervention. We will need to find a way to ensure we protect all intellectual property and proprietary information before we develop a plan to share IPD.

REFERENCES:
- [Background] Newlon JL, Campi JA, Rafie S, Meredith AH. Determining user implementation needs for pharmacist-prescribed contraception using concept mapping: A participatory, multiple stakeholder approach. Explor Res Clin Soc Pharm. 2024 Oct 11;16:100525. doi: 10.1016/j.rcsop.2024.100525. eCollection 2024 Dec. PMID 39512515
- [Background] Campi JA, Rafie S, Newlon JL, Meredith AH. Implementation of pharmacist-prescribed contraceptive services: A case series of early adopters. JAPhA Pract Innov. 2024 Jul;1(3):100011. doi: 10.1016/j.japhpi.2024.100011. Epub 2024 Apr 20. PMID 39420991